CLINICAL TRIAL: NCT05357118
Title: Battling Stigma for Service Engagement Among Women With HIV in Vietnam
Brief Title: Stigma Among Women With HIV in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Hanoi Medical University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Chunqing Lin, PhD, Assistant Professor-in-Residence, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1191; R21TW012018 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-05-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stigma, Social; HIV Infections; Discrimination, Sex
Keywords: Vietnam; Stigma; HIV; Women
MeSH Terms: conditions — Social Stigma; HIV Infections; Sexism

STUDY DESIGN:
Intervention Model Description: Women living with HIV/AIDS (WLHA) will attend an initial group preparation session in Month 1 to form a network with peers and prepare for the following online support groups. During Month 2-4, study investigators will teach cognitive, emotional, and behavioral strategies to cope with stigma and utilize social support to seek healthcare services through online group activities. During Month 4-6, WLHA will self-administer the online support groups without the intervention of study investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One arm (Experimental): The study is an one-arm pre- and post-design.
  Interventions: Behavioral: Suppress Stigma, Support Services

INTERVENTIONS:
Behavioral: Suppress Stigma, Support Services — Women living with HIV/AIDS (WLHA) will attend an initial group preparation session in Month 1 to form a network with peers and prepare for the following online support groups. During Month 2-4, study investigators will teach cognitive, emotional, and behavioral strategies to cope with stigma and utilize social support to seek healthcare services through online group activities. During Month 4-6, WLHA will self-administer the online support groups without the intervention of study investigators

SUMMARY:
Women living with HIV/AIDS (WLHA) bear a higher level of stigma because of their socio-cultural vulnerabilities. Women are more likely to internalize social stigma and produce a sense of shame and loss of self-worth, which results in a delay in health service seeking and compromised health outcomes. In Vietnam, stigma towards WLHA is exacerbated by the deeply rooted female inferiority. However, research targeting WLHA is generally lacking. We propose this study to address stigma among WLHA and explore the use of virtual support system in WLHA's service engagement in Vietnam. The 2-year study will proceed in two phases in Hanoi, Vietnam. Phase 1 will be formative studies, including in-depth interviews with 30 WLHA and focus groups with 20 service providers and community stakeholders. This phase aims to investigate the cultural and contextual background of HIV and gender roles in Vietnam and to identify effective strategies to support and engage WLHA in healthcare. These formative findings will inform the development of an intervention to be pilot tested in the next phase. Phase 2 will be a 6-month intervention pilot with 90 WLHA using an online/offline hybrid approach. During Month 1 of the pilot, WLHA will participate in an in-person section to form mutual support groups and prepare for the following online components. During Month 2-4 of the pilot, study investigators will teach WLHA a series of empowerment strategies to cope with stigma and utilize social support to seek healthcare services. These skills will be taught via interactive online group activities. During Month 4-6, WLHA will self-administer the online groups without the intervention of study investigators. WLHA's multidimensional stigma measures, mental health burdens, and service use self-efficacy will be assessed at baseline, month 4, and month 6. Progress data of the intervention will be documented to inform the feasibility and sustainability of the online support approach. Acceptability data and feedback will be collected from the WLHA participants upon completion of the 6-month pilot period.

DETAILED DESCRIPTION:
Women living with HIV/AIDS (WLHA) bear HIV stigma layered with gender disparity. They continue to suffer from internalized shame, which compromises their mental health and discourages them from seeking healthcare. Stigma among WLHA has the most detrimental impact on WLHA in Asian Countries, such as Vietnam, due to the deeply rooted male supremacy in the culture. The objective of this study is to investigate Vietnamese WLHA's cognitive, emotional, and behavioral responses to stigma, and test strategies to address the adverse impact of stigma on WLHA's health and service seeking. This proposed 2-year study, which will be conducted in Hanoi, Vietnam, will proceed in two phases.

In Phase 1, we will conduct formative studies, including in-depth interviews with 30 WLHA, one focus group with 10 healthcare providers, and one focus group with 10 community stakeholders. The aim of the formative study is to explore the cultural and contextual background of HIV stigma and gender disparity in Vietnam, investigate WLHA's barriers to access healthcare, identify locally available resources to combat stigma, and solicit feedback on some of the potential stigma-reduction intervention strategies. Phase 1 findings will inform the strategies to be pilot tested in Phase 2.

In Phase 2, the intervention will be piloted among 90 WLHA. The WLHA participants will be recruited from HIV testing sites, HIV outpatient clinics, obstetrics/maternity clinics, community-based organizations, and women's associations in Hanoi. The pilot testing period will be approximately six months. During the first month (Month 1), the WLHA will attend a group session to build initial contact with each other and prepare for the following online activities. During the preparation session, online support groups will be established using popular local socializing applications (e.g., Facebook). There will be approximately 30 WLHA in each online group. During the following three months (Month 2-4), study investigators will deliver stigma reduction intervention in the online groups, with focuses to address cognitive process of societal stigma, adjust negative emotional responses to stigma, and promote positive coping and active services seeking. During the final two months (Month 5-6), WLHA will continue the discussion and mutual support activities in the online groups without the intervention of study investigators. The online discussions will serve as process data to inform the usability and sustainability of the intervention. WLHA participants will be surveyed at baseline, 4-, and 6-month to assess their cognitive, emotional, behavioral responses to stigma, perceived social support, service utilization, and physical/mental health. In addition, final focus groups will be organized with participating WLHA to collect feasibility/acceptability evaluations and feedback for intervention components. The information will be used to refine the intervention and its implementation plan.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* being female at birth and currently
* being HIV-seropositive
* currently living in Hanoi and having no plan to move out of the area in the next six months
* have the cognitive capacity to participate in study activities as judged by the study recruiter

Exclusion Criteria:

* have been involved in intervention development activities
* inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Born as a female
Enrollment: 91 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Change in stigma | Baseline to 6-month
  The change in a scale to measure how WLHA's awareness of HIV stigma, agreement with stigma, coping with stigma. The items of the stigma measure are adopted based on Corrigan PW's Toolkit for Evaluating Programs Meant to Erase the Stigma of Mental Illness. (2008)

SECONDARY OUTCOMES:
Change in social support | Baseline to 6-month
  The change in social support measure appraisal support, informational support, emotional support, and spiritual support. The UCLA Social Support Inventory will be used (Schwarzer R, Dunkel-Schetter C, Kemeny M. The multidimensional nature of received social support in gay men at risk of HIV infection and AIDS. Am J Community Psychol. 1994 Jun;22(3):319-39. doi: 10.1007/BF02506869). Range 16-80, higher score indicates higher level of perceived social support.
Change in self-efficacy to tackle stigma and seek healthcare/social services | Baseline to 6-month
  The change in self-efficacy measure evaluates WLHA's level of confidence to tackle stigma and seek healthcare/social services, measured using the HIV Self-Efficacy (HIV-SE) scale developed by Shively and colleagues (Shively M, Smith T, Bormann J, Gifford A. Evaluating self-efficacy for HIV disease management skills. AIDS Behav. 2002;6:371-379. doi: 10.1023/A:1021156914683). The scale contains six domains including managing mood, managing medications, managing symptoms, managing fatigue, communicating with the healthcare provider, and getting support (Range 18-180, a higher score indicates a higher level of self-efficacy to tackle stigma and seek care).
Change in access to care | Baseline to 6-month
  The change in a measure evaluate WLHA's access to antiretroviral therapy and treatment for other comorbidities, adhering to medications, managing symptoms, and communicating with service providers, measured using the Barriers to Access to Care Evaluation scale (BACE; Clement, S., Brohan, E., Jeffery, D., Henderson, C., Hatch, S. L., & Thornicroft, G. (2012). Development and psychometric properties the Barriers to Access to Care Evaluation scale (BACE) related to people with mental ill health. BMC psychiatry, 12(1), 36). Range 12-48, higher score indicates higher barriers to access to treatment and care.
Change in health status | Baseline to 6-month
  The change in to measure evaluates WLHA's multidimensional health status, including physical health, physical functioning, mental health, and social functioning, measured with the SF-12 Health Survey (79. Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID: 8628042). Range 0-100; higher score indicates better physical and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers